CLINICAL TRIAL: NCT00134953
Title: Efficacy and Safety of Rivastigmine in Patients With Mild Cognitive Impairment
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Principal Investigator left the clinic and there was no one who could take over this study.
Sponsor: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CENA713BDE05
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2007-12-17 (Estimated); Status verified 2007-12

CONDITIONS: Cognitive Symptoms
Keywords: Mild cognitive impairment; Alzheimer's disease; Dementia; Mild Cognitive Impairment (MCI)
MeSH Terms: conditions — Neurobehavioral Manifestations; Cognitive Dysfunction; Alzheimer Disease; Dementia | interventions — Rivastigmine

INTERVENTIONS:
Drug: Rivastigmine

SUMMARY:
This study is designed to investigate the efficacy and safety of rivastigmine compared with placebo in patients with mild cognitive impairment (MCI).

ELIGIBILITY:
Inclusion Criteria:

* Males or females who are one year post-menopausal or without childbearing potential
* Between the ages of 50 and 85 years old
* Mild cognitive impairment confirmed by Mini Mental State Examination (MMSE) score between 23 and 27
* Cooperative, able to ingest oral medication, and able to complete all aspects of the study and capable of doing so, either alone or with the aid of a responsible caregiver, according to the investigator's judgement

Exclusion Criteria:

* A current diagnosis of cerebrovascular disease, any primary neurodegenerative disorder, or any other causes of neuropsychologic disturbances or secondary dementia
* A current diagnosis of epilepsy or depression, or any other diagnosis that may interfere with the patient's response to study medication
* An advanced, severe or unstable disease of any type that may interfere with efficacy evaluations

Other protocol-defined exclusion criteria may apply.

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2003-01; Study Completion 2004-05 (Actual)

PRIMARY OUTCOMES:
16 week's treatment with rivastigmine on alertness, memory, attention, cognitive flexibility, orientation and language in patients with mild cognitive impairment

SECONDARY OUTCOMES:
Safety of 16 week's treatment with rivastigmine in patients with mild cognitive impairment

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals Corporation, Study Director — Novartis Pharmaceuticals